CLINICAL TRIAL: NCT01470131
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled, 2-parallel Group, Phase 3 Study to Compare Efficacy and Safety of Masitinib 6 mg/kg/Day in Combination With Bortezomib and Dexamethasone to Placebo in Combination With Bortezomib and Dexamethasone in the Treatment of Patients With Relapsing Multiple Myeloma Who Received One Previous Therapy
Brief Title: A Phase 3 Study to Evaluate Efficacy and Safety of Masitinib in Patients With Relapse or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB06002
Record Dates: First submitted 2011-10-25; First posted 2011-11-11 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; relapse; second line therapy; bortezomib; dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — masitinib; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib (Experimental): Masitinib (6 mg/kg/day) in combination with Bortezomib and Dexamethasone
  Interventions: Drug: Masitinib; Drug: Bortezomib; Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo in combination with Bortezomib and Dexamethasone
  Interventions: Drug: Placebo; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Masitinib — Masitinib 6 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib
Drug: Placebo — Matching placebo
  Arms: Placebo
Drug: Bortezomib — Standard therapy (cycles of bortezomib)
  Other Names: Velcade
Drug: Dexamethasone — Standard therapy (cycles of dexamethasone)
  Other Names: Dexasone

SUMMARY:
The purpose of the study is to compare the efficacy and safety of masitinib 6 mg/kg/day in combination with bortezomib and dexamethasone to placebo in combination with bortezomib and dexamethasone in the treatment of patients with relapsing multiple myeloma who have received one previous therapy.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled, 2-parallel group, phase 3 study to compare efficacy and safety of masitinib 9 mg/kg/day to placebo in the treatment of patients with relapsing multiple myeloma who received one previous therapy.

Patients will receive study treatment (masitinib/placebo) with the standard therapy (bortezomib and dexamethazone).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with confirmed multiple myeloma requiring systemic therapy. A
2. Patient with multiple myeloma relapsing according to the International uniform response criteria for multiple myeloma (IMWG 2009/ revised Bladé criteria) to one previous line of treatment
3. Patient with measurable progressive disease

Exclusion Criteria:

1. Patient with peripheral neuropathy Grade >2
2. Patient with hypersensitivity to bortezomib, boron or dexamethasone
3. Patient whose disease progressed during or within 60 days of bortezomib treatment or of any other Multiple Myeloma therapy
4. Patient who received bortezomib within 6 months of randomization to this study
5. Past discontinuation of bortezomib due to associated grade 3 or higher adverse event
6. Patient with contra-indication to high dose of steroids (including ongoing active infection, use of live vaccines, virosis such as hepatitis, herpes, varicella, herpes zoster)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Analysis to be conducted after a minimum of 201 events

SECONDARY OUTCOMES:
Overall Time to Progression | time from the date of randomization to the date of documented progression during the study
Overall Survival | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Arnulf, MD, Principal Investigator — Hôpital Saint-Louis, Paris - France
Locations (13):
- United States (5):
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Carolinas Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Froedtert & Medical College of Wisconsin-CLCC, Milwaukee, Wisconsin
- France (8):
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CH Le Mans, Le Mans
  - Hôpital Universitaire Dupuytren, Limoges
  - Hôpital Ambroise Paré, Marseille
  - Hôpital de l'Hôtel Dieu, Nantes
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Saint Jean, Perpignan